CLINICAL TRIAL: NCT01745666
Title: Comparison Between Epinephrine and Exercise Test in QT Long Syndrome Patients With KCNQ1 or KCNH2 Mutation Without Long QT Interval in Rest ECG
Brief Title: Comparison Between Epinephrine and Exercise Test in QT Long Syndrome Patients
Acronym: QT long
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC11_0160
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Long QT Syndrome Type 1 or 2
Keywords: Long QT syndrome, stress tests
MeSH Terms: conditions — Romano-Ward Syndrome; Long QT Syndrome | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with KCNQ1 or KCNH2 mutation (Experimental)
  Interventions: Other: exercise test; Other: Epinephrine test
- patients WITHOUT KCNQ1 or KCNH2 mutation (control group) (Other)
  Interventions: Other: exercise test; Other: Epinephrine test

INTERVENTIONS:
Other: exercise test — Exercise test : Bruce protocol : exercise during 7 minutes, and rest during 6 minutes with registering of the electrocardiograms.
Other: Epinephrine test — Epinephrine test : 1 hour after exercise test : epinephrine infusion during 20 minutes, and monitoring during 30 minutes after stop infusion with registering of electrocardiograms.

SUMMARY:
The aim of the study is to evaluate the best stress exam to unmask long QT in patient with KCNQ1 or KCNH2 mutation without long QT interval in rest electrocardiogram.

DETAILED DESCRIPTION:
65 patients with KCNQ1 or KCNH2 mutation presenting QTc interval <470msec and 65 patients without KCNQ1 or KCNH2 mutation presenting QTc interval <470msec will be included.

All patients will have the 2 tests: exercise test and epinephrine test, in one half day.

At the end of the inclusions, two experts will examine examens results without knowing in which arm (mutated or not) the patient belongs.

ELIGIBILITY:
Inclusion Criteria:

Patients with QTc<470 msec, and with molecular analysis (KCNQ1 or KCNH2 genes) performed in order to include 65 patients with KCNQ1 or KCNH2 mutation and 65 patients without KCNQ1 or KCNH2 mutation (controls).

Exclusion Criteria:

* QTc interval >470msec
* Treatment interfering with cardiac repolarisation
* Under 15 years old
* Pregnant women
* Contraindication to exercise or epinephrine tests
* Patients without social coverage

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
to evaluate the best stress exam (exercise test OR epinephrine test)to unmask long QT syndrome. | day 1
  Exercise test and epinephrine test will be done at inclusion (day 1). The primary outcome of this study is to evaluate the best stress exam (exercise test versus epinephrine test), defined by a "positive" test to unmask long QT syndrome. Test is positive when QT interval lengthens 30 ms At the end of study inclusions, two reviewers will analyse, independently, electrocardiograms resulting from these tests to determine for each patient if a test was positive and which one. These reviewers will do this job without being informed of the patient status (mutated patient or not mutated patient (control)).

SECONDARY OUTCOMES:
to evaluate each test characteristics | Day 1
  Exercise test and epinephrine test will be done at inclusion (day 1). The secondary outcome is to evaluate each test (exercise test and epinephrine test) characteristics. At the end of study inclusions, two reviewers will independently analyse electrocardiograms resulting from these tests to evaluate their characteristics.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Bordeaux Universitary Hospital, Bordeaux
  - Marseille Universitary Hospital, Marseille
  - CHU Montpellier, Montpellier
  - Nantes Universitary Hospital, Nantes
  - Rennes Universitary Hospital, Rennes
  - CHU Rouen, Rouen
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours